CLINICAL TRIAL: NCT03736070
Title: Assessment of Routine Oral Screening Programs for New Prisoners in France
Brief Title: Assessment of Routine Oral Screening Programs for New Prisoners
Acronym: DepiDent
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: General Health Office, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0069
Record Dates: First submitted 2018-02-01; First posted 2018-11-08 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Oral Disease
MeSH Terms: conditions — Mouth Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2018, 10 detention centers in France will start organisational programs to improve the quality of screening of oral diseases, relatively to French recommendations, among new prisoners in France. Our study aims 1) to assess the prevalence and nosology of oral diseases ; 2) to describe the care pathway of participants during their stay in the detention center where they were included ; 3) to assess the cost of care per patient, from a societal perspective, using a top-down method.

ELIGIBILITY:
Inclusion criteria:

* new prisoners
* fluent French language

Exclusion criteria:

* adult guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: New prisoners
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Description of the oral problems of people entering detention | 1 day
  Description of the oral problems of people entering detention : Any oral disease at inclusion (prevalence study)

SECONDARY OUTCOMES:
attending to consultations | The collection of data will end at the discharge of the participant, or at 6 months after inclusion.
  attending to consultations : The rate of attended visits is defined as the number of visits attended by the patient, divided by the number of scheduled visits, during the prison stay of the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Claire M DUFLOS, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC